CLINICAL TRIAL: NCT06022952
Title: Randomized, Single Center Controlled Trial of the Effect of the "Stone MD" Mobile App on the Prevention of Forgotten Ureteral Stents in Patients With Urolithiasis
Brief Title: The Impact of the "Stone MD" Mobile App on the Prevention of Forgotten Ureteral Stents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Stone_MD_forgotten_stent
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients who have used the Stone MD mobile app
  Interventions: Other: Stone MD stent radar
- Group B (Active Comparator): Patients who have not used the Stone MD mobile app
  Interventions: Other: Stone MD stent radar

INTERVENTIONS:
Other: Stone MD stent radar — Mobile app

SUMMARY:
The Impact of the "Stone MD" Mobile App on the Prevention of Forgotten Ureteral Stents

DETAILED DESCRIPTION:
Inclusion Criteria:

1. Male and female patients aged 18 to 80 years who have a Ch 4.7-6.0 polyurethane ureteral stent

Exclusion Criteria:

1. Active phase of urinary tract infection
2. Insufficient level of social adaptation
3. The patient does not have a smartphone with Internet access

All patients will be randomized into 2 groups:

* group A - patients who used the Stone MD mobile application
* group B - patients who did not use the mobile application Patients are to be assigned a randomization number that will match their treatment. Block randomization using 10 blocks is to be performed by a central randomization organization (www.randomize.net) using a computerized algorithm.

"Stent Radar" - part of the "Stone MD" mobile application. This tool is designed for the patient to remove the ureteral stent using a mobile application within the time period prescribed by the doctor. After the operation, the patient independently enters the data related to the installation of the stent in the Stent Radar section of the Stone MD mobile application. This data includes: the name of the stent, the side of insertion, and the estimated date of removal. In a few days, a push notification appears in the application stating that it is necessary to consult a doctor for the timely removal of the stent. Thus, it is almost impossible to forget to remove the stent.

At discharge, we strongly recommend that all patients install the Stone MD mobile app on their smartphone. In the postoperative period, all patients will be monitored. In the event that 2 weeks after the expected date of removal, the patient does not get in touch, he will receive a call from the clinic, reminding him of the necessary visit (to remove the stent).

Primary assessed outcomes:

1. Number of patients who removed the stent on time in both groups
2. Number of patients who delayed stent removal in both groups (less than 14 days)
3. Number of patients who forgot to remove the stent in both groups (removed the stent more than 14 days from the expected date of removal)

Secondary assessed outcomes:

1. Assessment of Stone-free status after surgery by performing computed tomography of kidneys and urinary tract without intravenous contrasting 1 month after surgery

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 to 80 years who have a Ch 4.7-6.0 polyurethane ureteral stent

Exclusion Criteria:

1. Active phase of urinary tract infection
2. Insufficient level of social adaptation
3. The patient does not have a smartphone with Internet access

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Removed on time | 30 days
  Number of patients who removed the stent on time in both groups
Delayed stent removal | 30 days
  Number of patients who delayed stent removal in both groups (less than 14 days)
Forgotten stent removal | 30 days
  Number of patients who forgot to remove the stent in both groups (removed the stent more than 14 days from the expected date of removal)

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - First Pavlov Saint Petersburg University, Saint Petersburg
  - Saint Petersburg State University Hospital, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Undecided